CLINICAL TRIAL: NCT04112329
Title: Effects of 8 Weeks of High-intensity Exergaming on Cardiorespiratory Fitness and Physical Activity Levels in Sedentary Adults
Brief Title: Exergaming for Better Physical Fitness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019/1083
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Sedentary Lifestyle
Keywords: Exercise therapy; Physical fitness; Gaming; Child; Healthy lifestyle; Fitness testing
MeSH Terms: conditions — Sedentary Behavior | interventions — Exergaming

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergaming (Experimental): Will use the PlayPulse exergame for 45 minutes a minimum of two times per week for 8 weeks
  Interventions: Behavioral: Exergaming
- Control (No Intervention): Asked to continue with their normal daily routine

INTERVENTIONS:
Behavioral: Exergaming — will use the PlayPulse exergame for 45 minutes a minimum of two times per week for 8 weeks.
  Arms: Exergaming

SUMMARY:
The purpose of this project is to assess if playing a newly developed videogame that require physical activity (e.g. exergame) can lead to increased physical activity, aerobic fitness and health benefits in sedentary adults. The project will include 28 sedentary adults, 18 years and above, who are not sufficiently active according to current guidelines defined as doing (<150 minutes/week of moderate intensity physical activity or <75 minutes/week of vigorous physical activity and/or do not do any regular endurance training ). The physical fitness (maximal oxygen consumption), blood pressure, body composition and objectively measured physical activity will be tested before and after the intervention period.

Also, the participants gaming frequency will be registered throughout the 8 week period. Aim of this study is to investigate if access to this game can provide health benefits for adults who are not motivated to take part in regular physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (<150 mins of moderate intensity physical activity/week) and/or do not regularly take part in endurance training.
* Able to ride a bike for up to 60 minutes

Exclusion Criteria:

* Known cardiovascular disease
* Taking beta-blockers or anti-arrhythmic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
VO2max (Maximal Aerobic Capacity) | 8 weeks

SECONDARY OUTCOMES:
Daily average energy expenditure | 8 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period and after intervention period (8 weeks).
Daily average number of steps | 8 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period and after intervention period (8 weeks).
Daily time in sedentary activity (< 3.0 metabolic equivalents = METs) | 8 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period and after intervention period (8 weeks).
Daily time in moderate intensity activity (3.0-6.0 metabolic equivalents = METs) | 8 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period and after intervention period (8 weeks).
Daily time in vigorous intensity activity (6.0-9.0 metabolic equivalents = METs) | 8 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period and after intervention period (8 weeks).
Daily time in very vigorous intensity activity (>9.0 metabolic equivalents = METs) | 8 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period and after intervention period (8 weeks).
Daily average total physical activity duration | 8 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period and after intervention period (8 weeks).
Bioelectrical impedance | 8 weeks
  Measured by activity monitors (SenseWear Armband) which participants will wear for one week at start of intervention period and after intervention period (weeks).
Blood Pressure | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, Study Director — Norwegian University of Science and Technology; Trine Moholdt, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Medical Imaging, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Berg J, Haugen G, Wang AI, Moholdt T. High-intensity exergaming for improved cardiorespiratory fitness: A randomised, controlled trial. Eur J Sport Sci. 2022 Jun;22(6):867-876. doi: 10.1080/17461391.2021.1921852. Epub 2021 May 16. PMID 33944698